CLINICAL TRIAL: NCT07286968
Title: Gastro-Intestinal Digestion and Physiology After Bariatric Surgery
Acronym: GIBa
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S70844; CIV-25-08-054154 (Other: AFMPS - FAGG)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Surgery; Roux-en Y Gastric Bypass; Sleeve Gastrectomy; Obesity & Overweight
Keywords: Gastro-intestinal aspiration; ingestible telemetric capsule
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Roux-en-Y gastric bypass: Patients who had undergone Roux-en-Y gastric bypass surgery
  Interventions: Other: Gastro-intestinal aspiration; Device: Telemetric
- Sleeve gastrectomy: Patients who had undergone sleeve gastrectomy surgery
  Interventions: Other: Gastro-intestinal aspiration; Device: Telemetric
- Patients living with obesity: Patients without previous bariatric surgery
  Interventions: Other: Gastro-intestinal aspiration; Device: Telemetric

INTERVENTIONS:
Other: Gastro-intestinal aspiration — Aspiration of fluids from the stomach and small intestine using a naso-intestinal catheter.
Device: Telemetric — Telemetric ingestible capsule

SUMMARY:
The goal of this clinical trial is to characterize gastrointestinal digestion and physiology in patients after bariatric surgery, or people living with obesity. The main question it aims to answer is: what is the status of gastrointestinal digestion and physiology after bariatric surgery? Participants will have two study visits: 1) participants will undergo collection of gastrointestinal samples and 2) participants will ingest an ingestible capsule that measures multiple physiological parameters along the gastrointestinal tract.

DETAILED DESCRIPTION:
This clinical trial aims to characterize gastric and pancreatic enzyme activity in adults aged 18 to 65 who have previously (at least 1 year ago) undergone Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG), as well as in individuals with obesity. In addition, the study seeks to quantify bile acid concentrations and pH at various locations within the gastrointestinal tract and to assess gastrointestinal transit time. During the study, aspirates will be collected from multiple regions of the gastrointestinal tract using a naso-intestinal catheter (study visit 1). An ingestible capsule will also be used to obtain continuous in vivo measurements of physiological conditions along the entire gastrointestinal tract (study visit 2).

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this Investigation have to meet all of the following criteria:

1. Voluntary written informed consent of the participant has been obtained prior to any screening procedures
2. Age: 18-65 years

   Specific inclusion criteria for the different patient populations:

   Patients with obesity:
3. Body Mass Index: > 30 kg/m2

   Patients after bariatric surgery:
4. Surgery: at least one year after Roux-en-Y gastric bypass or sleeve gastrectomy

Exclusion Criteria:

Participants eligible for this Investigation must not meet any of the following criteria:

1. Patient has history of more than one bariatric surgery
2. Patient has a waist circumference > 125.6 cm
3. Patient had gastrointestinal surgery in the past three months
4. Patient has a pacemaker, defibrillator, infusion pump, or other portable or implanted electromedical device
5. Patient had frequent exposure to X-rays in the past year
6. Patient has swallowing disorders, among others: dysphagia for food or pills, any oropharyngeal or oesophageal stricture, anxiety or functional abnormality
7. Patient has Crohn's disease or Diverticulitis
8. Patient has gastrointestinal strictures, fistulas or physiological/mechanical obstructions
9. Patient has gastric bezoar
10. Patient has a history of complex bowel resection or known abdominal adhesions
11. Patient has short bowel syndrome or ostomy
12. Patient has currently ongoing infections
13. Patient is planned to undergo usage of rectal foam/enema or treatment with adjuvant chemotherapy or radiotherapy
14. Patient is currently on parenteral diet
15. Patient is planned to undergo MRI procedure during usage of the wireless capsule
16. Patient is working in a professional healthcare facility (e.g. hospital, dental office, emergency room), military area (e.g. submarine, near radar installation), or heavy industrial area (e.g. power plants, automotive, mining, refineries) during the duration of the clinical investigation
17. Patient is pregnant, breastfeeding, actively trying to get pregnant or had recent childbirth in last 6 months
18. Patient cannot discontinue medication that affects gastrointestinal transit time and/or pH for at least 3 days before and during the study (and 4 weeks for weekly/long-acting GLP-1 analogues such as Saxenda, Ozempic, Wegovy, Mounjaro). This includes opioids (e.g., morphine, codeine), proton pump inhibitors (e.g., omeprazole, esomeprazole, pantoprazole), H2-receptor antagonists (e.g., cimetidine, famotidine), antacids, sucralfate, prokinetics (e.g., domperidone, metoclopramide), antidiarrheal agents (e.g., loperamide), antibiotics, probiotics and prebiotics.
19. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CIP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously undergone a RYGB surgery, SG surgery, or people with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Activity of gastric lipase | 2 hours
  Gastric pouch and sleeve samples will be analysed for gastric lipase activity (described in U)
Activity of pepsin | 2 hours
  Gastric pouch and sleeve samples will be analysed for pepsin activity (described in U)
Activity of trypsin | 2 hours
  Samples collected in the duodenum and jejunum; or roux- and common-limb will be analysed for trypsin activity (described in U).
Activity of chymotrypsin | 2 hours
  Samples collected in the duodenum and jejunum; or roux- and common-limb will be analysed for chymotrypsin activity (described in U).
Activity of α-amylase | 2 hours
  Samples collected in the duodenum and jejunum; or roux- and common-limb will be analysed for α-amylase activity (described in U).
Activity of pancreatic lipase | 2 hours
  Samples collected in the duodenum and jejunum; or roux- and common-limb will be analysed for pancreatic lipase activity (described in U).

SECONDARY OUTCOMES:
Concentration of total bile acids | 2 hours
  The total bile acid concentrations will be measured in all samples
pH | 2 hours
  pH will be measured in all gastro-intestinal samples
Total transit time | 48 hours
  Total transit time will be measured by the GISMO GEN I ingestible sensor (described in minutes).
Gastric emptying time | 48 hours
  Gastric emptying time will be measured by the GISMO GEN I ingestible sensor (described in minutes).
Small intestinal transit time | 48 hours
  Small intestinal transit time will be measured by the GISMO GEN I ingestible sensor (described in minutes).
Large intestinal transit time | 48 hours
  Large intestinal transit time will be measured by the GISMO GEN I ingestible sensor (described in minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided